CLINICAL TRIAL: NCT04761237
Title: A Research of Central Venous-arterial Carbon Dioxide Difference Has Guiding Significance for Severely Burn Patients in Liquid Resuscitation During Early Escharectomy
Brief Title: The Value of Central Venous-arterial Carbon Dioxide Difference
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Liang Bing (Other)
Responsible Party: Sponsor-Investigator, Liang Bing, Associate chief physician, Guangzhou Red Cross Hospital
Organization: Guangzhou Red Cross Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2015-047-01
Record Dates: First submitted 2021-01-19; First posted 2021-02-18 (Actual); Last update posted 2021-02-18 (Actual); Status verified 2021-02

CONDITIONS: Jugular Veins; Radial Artery; Carbon Dioxide
Keywords: central venous-arterial carbon dioxide difference; liquid resuscitation; tissue perfusion and oxygenation

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants are prevented from having knowledge of the interventions assigned to individual participants.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): (H-P) : Pcv-aCO2≥6mmHg between T base and T 0h.;
  Interventions: Drug: Goal-directed fluid therapy (GDET)
- Group 2 (Experimental): (L-P) : Pcv-aco2< 6mmHg at T base and≥6mmHg at T 0h
  Interventions: Drug: Goal-directed fluid therapy (GDET)

INTERVENTIONS:
Drug: Goal-directed fluid therapy (GDET) — Compensatory dilatation was performed firstly and 5ml/kg crystal solution was added within 30min before induction of anesthesia.When SVV≥13%, infusion of colloidal solution 2ml/kg was performed 15-20 minutes.If the increase of SV was≥10% after the liquid impact and the SVV was still≥13%, the colloidal solution was used again for 2mL/kg and the infusion was maintained until the SVV < 13%.The infusion was stopped when the SVV < 10%.If the increase of SV was less than 10% or CI < 2.0L/min/m2 after infusion, dobutamine was given intravenously to observe the change of SV. If the increase of SV was greater than 10%, dobutamine could be maintained and the above fluid regimen continued.If the increase of SV was less than 10% and MAP≥65mmHg, the infusion of liquid was stopped and replaced with 4ml/kg/h infusion for maintenance.If the increase of SV was less than 10% and MAP was less than 65mmHg, the infusion was suspended.

SUMMARY:
By observing the changes of Central venous-arterial partial pressure difference of carbon dioxide [P (v-a) CO2] in liquid resuscitation during early escharectomy in patients with large-scale burns, We investigate the effect of P (v-a) CO2 on postoperative tissue perfusion and oxygenation in order to seek a more effective intergrated target plan of liquid resuscitation for burn patients.

DETAILED DESCRIPTION:
Objective: By observing the changes of Central venous-arterial partial pressure difference of carbon dioxide [P (v-a) CO2] in liquid resuscitation during early escharectomy in patients with large-scale burns, We investigate the effect of P (v-a) CO2 on postoperative tissue perfusion and oxygenation in order to seek a more effective intergrated target plan of liquid resuscitation for burn patients.

Methods: a prospective observational study was conducted on 145 patients with extensive burns admitted to surgical intensive care unit（SICU）of Guangzhou Red Cross hospital from January 2016 to December 2019. All patients received hemodynamic monitoring and goal-directed fluid therapy, patients with central venous oxygen saturation (ScvO2)< 70% were excluded. Patients were divided into the following groups according to the changing trend of Pcv-aCO2 between T base (before induction) and T 0h (after surgery) : group 1 (H-H) : Pcv-aCO2≥6mmHg between T base and T 0h. Group 2 (L-H) : Pcv-aco2< 6mmHg at T base and≥6mmHg at T 0h; Group 3 (H-L) : Pcv-aCO2≥6mmHg at T base and < 6mmHg at T 0h. Group 4( L-L) : Pcv-aCO2 < 6mmHg between T base and T0h.Postoperative basic physiological indicators such as heart rate（HR）, blood pressure, central venous pressure (CVP), cardiac output index (CI), Pcv-aCO2 and lactic acid were recorded at 0 and 18 hours after surgery. Oxygen dynamic indicators such as oxygen delivery index (DO2I), oxygen consumption index (VO2I), oxygen uptake rate (O2ER) and so on were calculated. Pearson correlation analysis was used to evaluate the correlation between Pcv-aCO2 and CI. The change of tissue perfusion and oxygenation with different levels of Pcv-aCO2 after fluid resuscitation were analyzed.

ELIGIBILITY:
Inclusion Criteria:

1. ASAI-II
2. New York Heart Association classification of cardiac function I-II
3. Estimated time of operation<3h
4. The circulatory system of patients is stable after thrapy：CVP8～12 mmHg；MAP≥65 mmHg；urine volume>0.5m1/kg/ h；ScvO2：≥70％。

Exclusion Criteria:

1. Anesthetic drug allergy or contraindication
2. Patients with cardiopulmonary system disease、cardiopulmonary function abnormality、severe inhalation injuryand severe visceral injury.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
Central venous oxygen saturation | From start anesthesia until end of anesthesia, up to a maximum of 6 hours
  Central venous oxygen saturation in venous blood
Lactic acid value | From start anesthesia until end of anesthesia, up to a maximum of 6 hours
  Lactic acid level in arterial blood